CLINICAL TRIAL: NCT00977925
Title: A Phase III Randomized, Controlled, Superiority Study Evaluating the Fibrin Pad Versus Standard of Care Treatment in Controlling Severe Soft Tissue Bleeding During Abdominal, Retroperitoneal, Pelvic, and Thoracic Surgery
Brief Title: The Severe Soft Tissue Bleeding Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 400-08-002
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Soft Tissue Bleeding
Keywords: Hemostasis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrin Pad (Experimental)
  Interventions: Biological: Fibrin Pad
- Standard of Care (Active Comparator)
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Biological: Fibrin Pad — Fibrin Pad is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
  Arms: Fibrin Pad
Procedure: Standard of Care — Standard of Care is a composite of techniques/methods typically used by the surgeon to control severe bleeding.
  Arms: Standard of Care

SUMMARY:
The objective of this study is to evaluate the safety and hemostatic effectiveness of the Fibrin Pad (FP) versus standard of care treatment (SoC) in controlling challenging severe soft tissue bleeding during abdominal, pelvic, retroperitoneal, and (non-cardiac) thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >= 18 years of age, requiring elective, open, abdominal, retroperitoneal, pelvic or thoracic (non-cardiac) surgical procedures;
* Presence of an appropriate severe bleeding soft tissue Target Bleeding Site (TBS) as identified intra-operatively by the surgeon;
* Subjects must be willing to participate in the study, and provide written informed consent.

Exclusion Criteria:

* Subjects with any intra-operative findings identified by the surgeon that may preclude conduct of the study procedure;
* Bleeding site is from large defects in arteries or veins where the injured vascular wall requires repair with maintenance of vessel patency and which would result in persistent exposure of the FP to blood flow and pressure during healing and absorption of the product;
* Subject with TBS within an actively infected field;
* Bleeding site is in, around, or in proximity to foramina in bone, or areas of bony confine;
* Subjects with known intolerance to blood products or to one of the components of the study product;
* Subjects unwilling to receive blood products;
* Subjects with known immunodeficiency diseases (including known HIV);
* Subjects who are known, current alcohol and / or drug abusers;
* Subjects who have participated in another investigational drug or device research study within 30 days of enrollment;
* Female subjects who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving hemostasis at the Target Bleeding Site. Hemostasis is defined as no detectable bleeding at the TBS. | Intra-operative

SECONDARY OUTCOMES:
Proportion of subjects achieving hemostatic success at 10 minutes following randomization | Intra-operative
Absolute time to hemostasis | Intra-operative
Proportion of subjects requiring re-treatment at the TBS prior to wound closure | Intra-operative
Incidence of treatment failures | Intra-operative
Incidence of adverse events that are potentially related to bleeding at the TBS | Intra-operative through 60 days
Incidence of adverse events that are potentially related to thrombotic events; | Intra-operative through 60 days
Incidence of adverse events | Intra-operative through 60 days

CONTACTS AND LOCATIONS:
Overall Officials: James Hart, MD, Study Director — Ethicon, Inc.
Locations (16):
- Australia (4):
  - Bankstown Hospital, Bankstown
  - Flinders Medical Centre, Bedford Park
  - The Townsville Hospital, Douglas
  - Royal Melbourne Hospital, Parkville
- Germany (4):
  - University Hospital of the University of Saarland, Homburg/Saar, Homburg/Saar
  - Department of Surgery, University of Heidelberg, Heidelberg
  - Krankenhaus Salem, Heidelberg
  - Vincentius-Klinken, Karlsruhe
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - North Shore Hospital, Auckland
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrookes Hospital, Cambridge
  - The Royal Infirmary of Edinburgh, Edinburgh
  - St. James University Hospital, Leeds
  - St Bartholomew's Hospital, London
  - Nottingham City Hospital, Nottingham

REFERENCES:
- [Result] Koea J, Baldwin P, Shen J, Patel B, Batiller J, Arnaud A, Hart J, Hammond J, Fischer C, James Garden O. Erratum to: Safety and Hemostatic Effectiveness of the Fibrin Pad for Severe Soft-Tissue Bleeding During Abdominal, Retroperitoneal, Pelvic, and Thoracic (Non-cardiac) Surgery: A Randomized, Controlled, Superiority Trial. World J Surg. 2015 Oct;39(10):2610. doi: 10.1007/s00268-015-3163-9. No abstract available. PMID 26216641
- [Result] Koea J, Baldwin P, Shen J, Patel B, Batiller J, Arnaud A, Hart J, Hammond J, Fischer C, James Garden O. Safety and Hemostatic Effectiveness of the Fibrin Pad for Severe Soft-Tissue Bleeding During Abdominal, Retroperitoneal, Pelvic, and Thoracic (Non-cardiac) Surgery: A Randomized, Controlled, Superiority Trial. World J Surg. 2015 Nov;39(11):2663-9. doi: 10.1007/s00268-015-3106-5. PMID 26041587
- [Derived] Corral M, Ferko N, Hollmann S, Hogan A, Jamous N, Batiller J, Shen J. Clinician reported ease of use for a novel fibrin sealant patch for hemostasis: results from four randomized controlled trials. Curr Med Res Opin. 2016;32(2):367-75. doi: 10.1185/03007995.2015.1128405. Epub 2015 Dec 21. PMID 26636489